CLINICAL TRIAL: NCT00728078
Title: Low-Dose Thalidomide as Adjuvant Therapy After Radiofrequency Ablation for Hepatocellular Carcinoma
Acronym: LDT-RFA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: cancer canter, Sun Yat-sen University, cancer canter, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFA005
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: hepatocellular carcinoma; liver cancer; radiofrequency ablation; thalidomide
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): low-dose thalidomide adjuvant therapy after RFA for HCC
  Interventions: Drug: thalidomide
- 2 (No Intervention): control group

INTERVENTIONS:
Drug: thalidomide — thalidomide 50mg tid for 6 months
  Arms: 1

SUMMARY:
The purpose of the investigators' study is to prospectively evaluate whether low-dose thalidomide adjuvant therapy will improve the outcome of radiofrequency ablation for hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
Our previous studies showed that radiofrequency ablation (RFA) was as effective as liver resection for small hepatocellular carcinoma (HCC), but the recurrence rates after RFA were relatively high. Adjuvant therapies maybe reduce the recurrence rate. Phase 1 and 2 studies showed that thalidomide was a safety and effective treatment for HCC, especially for small HCC with liver cirrhosis. So we proposed that low-dose thalidomide adjuvant therapy will improve the disease progress free survivals and overall survivals after RFA for HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years, who refused surgery or first recurrence after hepatectomy
* A solitary HCC 3.1-7.0cm in diameter, or 2-3 lesions, sums of diameters ≤ 7.0cm
* Lesions being visible on ultrasound (US) and with an acceptable/safe path between the lesion and the skin as shown on US
* No extrahepatic metastasis
* No imaging evidence of invasion into the major portal/hepatic vein branches
* No history of encephalopathy, ascites refractory to diuretics or variceal bleeding
* A platelet count of > 40,000/mm3
* No previous treatment of HCC except liver resection

Exclusion Criteria:

* Patient compliance is poor
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted
* History of cardiac disease:

  * congestive heart failure > New York Heart Association (NYHA) class 2
  * active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted)
  * cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, *calcium channel blocker or digoxin
  * uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of 3 antihypertensive drugs)
* Active clinically serious infections (> grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known Central Nervous System tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* Distantly extrahepatic metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
progress free survival | 1,3,5-year
morbility | one month

SECONDARY OUTCOMES:
overall survival | 1,3,5-year
recurrence rate | 1,3,5-year

CONTACTS AND LOCATIONS:
Overall Officials: min-shan chen, MD, Principal Investigator — Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Chen MS, Li JQ, Zheng Y, Guo RP, Liang HH, Zhang YQ, Lin XJ, Lau WY. A prospective randomized trial comparing percutaneous local ablative therapy and partial hepatectomy for small hepatocellular carcinoma. Ann Surg. 2006 Mar;243(3):321-8. doi: 10.1097/01.sla.0000201480.65519.b8. PMID 16495695
- [Result] Buscarini L, Buscarini E, Di Stasi M, Vallisa D, Quaretti P, Rocca A. Percutaneous radiofrequency ablation of small hepatocellular carcinoma: long-term results. Eur Radiol. 2001;11(6):914-21. doi: 10.1007/s003300000659. PMID 11419162